CLINICAL TRIAL: NCT02425150
Title: Treatment of Keratoconus With Advanced Corneal Crosslinking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Anders Behndig, Professor, Umeå University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRXL
Record Dates: First submitted 2015-04-13; First posted 2015-04-23 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Keratoconus
Keywords: Keratoconus; Corneal crosslinking; Corneal biomechanics; Corneal densitometry; Scheimpflug photography
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Corneal reshaping/crosslinking (CRXL) (Experimental): Corneal crosslinking with compression of the cornea using a sutured rigid contact lens during the treatment.
  Interventions: Procedure: Corneal reshaping/crosslinking (CRXL)
- Corneal crosslinking (CXL) (Active Comparator): Standard corneal crosslinking using the Dresden protocol.
  Interventions: Procedure: Corneal Crosslinking (CXL)
- Control group to CRXL (No Intervention): Healthy subjects, age- and sex-matched to the CRXL group.
- Control group to CXL (No Intervention): Healthy subjects, age- and sex-matched to the CXL group.

INTERVENTIONS:
Procedure: Corneal reshaping/crosslinking (CRXL) — The keratoconus cornea is treated with epithelial debridement in local anesthesia, is soaked in Riboflavin by repeated topical application during 30 minutes. A flat, rigid contact lens is sutured to the cornea and the cornea and is then irradiated with ultraviolet light 5.4 J/cm2 during 30 minutes.
  Arms: Corneal reshaping/crosslinking (CRXL)
Procedure: Corneal Crosslinking (CXL) — The keratoconus cornea is treated with epithelial debridement in local anesthesia, is soaked in Riboflavin by repeated topical application during 30 minutes. The cornea and is then irradiated with ultraviolet light 5.4 J/cm2 during 30 minutes.
  Arms: Corneal crosslinking (CXL)

SUMMARY:
The purpose of this study was to determine whether mechanical compression of the cornea during corneal crosslinking for keratoconus using a sutured rigid contact lens can improve the optical outcomes of the treatment.

DETAILED DESCRIPTION:
The study is designed as a prospective, open, randomized controlled trial involving patients aged 18-28 years of both genders with uni- or bilateral keratoconus planned for routine corneal crosslinking at the Department of Ophthalmology, Umeå University Hospital, Umeå, Sweden. The study involves 30+30 eyes with keratoconus, which are randomized to receive either conventional corneal crosslinking (n=30) using the Dresden protocol or a modified treatment - corneal reshaping and crosslinking (n=30), where a rigid contact lens is sutured to the cornea during the treatment to flatten the corneal curvature and potentially improve the optical outcome after the treatment. Patients are randomized utilizing a list of unique random numbers between 1 and 60. All patients are informed about the procedures before consenting to participate in the study. The study also involves 60 eyes of healthy age- and sex-matched control subjects.

At baseline, before treatment, each eye is evaluated with autorefractometer measurement, best spectacle-corrected LogMAR visual acuity, Pentacam Scheimpflug photography, Goldmann applanation tonometry and biomicroscopy. The corneal biomechanical characteristics are assessed with applanation resonance tonometry and the ocular response analyzer. The investigations are repeated at 1 month, 6 months, 2 years and 5 years after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for corneal crosslinking.
* Progressive keratoconus documented with Scheimpflug photography using the Pentacam Scheimflug camera and/or repeated subjective refraction and keratometry.
* A keratoconus diagnosis based on the Amsler-Krumeich grading and the "Total Deviation" KC quantification value from the "Belin-Ambrosio enhanced ectasia" measurements of the Pentacam Scheimpflug camera, and an altered red reflex and/or an irregular cornea seen as distortion of the keratometric mires.
* Minimum corneal thickness of 400 µm at the thinnest point after epithelial removal.
* 18-28 years of age
* No ocular abnormalities except keratoconus
* No previous ocular surgery
* No cognitive insufficiency interfering with the informed consent.

Exclusion Criteria:

* Age under 18 or over 28
* Any corneal abnormalities except keratoconus
* Previous ocular surgery
* Cognitive insufficiency.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2009-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in refraction | 1, 6, 24 and 60 months after the treatment
  Refractive errors, including lower and higher order aberrations in the cornea

SECONDARY OUTCOMES:
Change from baseline in ETDRS LogMAR visual acuity | 1, 6, 24 and 60 months after the treatment
  Uncorrected and best spectacle corrected visual acuity measured with the Early treatment diabetic retinopathy study, graded in logarithmic values of the minimal angle of resolution
Change from baseline in corneal biomechanical stability measured with ORA | 1, 6, 24 and 60 months after the treatment
  Biomechanical stability assessed with the ocular response analyzer
Change from baseline in corneal biomechanical stability measured with ART | 1, 6, 24 and 60 months after the treatment
  Biomechanical stability assessed with the applanation resonance tonometer
Change from baseline in corneal biomechanical stability measured with GAT | 1, 6, 24 and 60 months after the treatment
  Biomechanical stability assessed with the Goldmann applanation tonometer
Change from baseline in corneal densitometry | 1, 6, 24 and 60 months after the treatment
  Corneal light reflectivity (back scatter) assessed with the Pentacam HR Scheimpflug camera

CONTACTS AND LOCATIONS:
Overall Officials: Anders Behndig, Professor, Principal Investigator — Umeå University

REFERENCES:
- [Background] Beckman Rehnman J, Behndig A, Hallberg P, Linden C. Initial results from mechanical compression of the cornea during crosslinking for keratoconus. Acta Ophthalmol. 2014 Nov;92(7):644-9. doi: 10.1111/aos.12380. Epub 2014 Mar 15. PMID 24628999
- [Background] Beckman Rehnman J, Behndig A, Hallberg P, Linden C. Increased corneal hysteresis after corneal collagen crosslinking: a study based on applanation resonance technology. JAMA Ophthalmol. 2014 Dec;132(12):1426-32. doi: 10.1001/jamaophthalmol.2014.3029. PMID 25171564
- [Result] Beckman Rehnman J, Janbaz CC, Behndig A, Linden C. Spatial distribution of corneal light scattering after corneal collagen crosslinking. J Cataract Refract Surg. 2011 Nov;37(11):1939-44. doi: 10.1016/j.jcrs.2011.05.028. Epub 2011 Aug 27. PMID 21873026
- [Derived] Rehnman JB, Linden C, Hallberg P, Behndig A. Treatment Effect and Corneal Light Scattering With 2 Corneal Cross-linking Protocols: A Randomized Clinical Trial. JAMA Ophthalmol. 2015 Nov;133(11):1254-60. doi: 10.1001/jamaophthalmol.2015.2852. PMID 26312777